CLINICAL TRIAL: NCT01634529
Title: A Double-blind, Randomised, Placebo-controlled Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Ascending Oral Doses of V158866 in Healthy Volunteers
Brief Title: Single and Multiple Ascending Dose Study of V158866 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vernalis (R&D) Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: V158866-1Pa-01
Record Dates: First submitted 2011-07-21; First posted 2012-07-06 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: First in Man Study

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single Ascending Dose (Experimental): Single ascending doses of V158866 compared to Placebo
  Interventions: Drug: V158866
- Multiple ascending doses (Experimental): Multiple ascending doses of V158866 compared to Placebo
  Interventions: Drug: V158866

INTERVENTIONS:
Drug: V158866 — Single ascending oral doses of V158866 and Placebo
  Arms: Single Ascending Dose
Drug: V158866 — Multiple ascending oral doses of V158866 and Placebo
  Arms: Multiple ascending doses

SUMMARY:
The purpose of this study is to investigate whether V158866 is safe when given to healthy male subjects in single and multiple doses.

DETAILED DESCRIPTION:
A first in human study:

To evaluate the safety and tolerability of single and multiple doses of V158866 in healthy male subjects To assess the pharmacokinetics (PK) of V158866 in healthy male subjects To assess the pharmacodynamics (PD) of V158866 by determining whether V158866 inhibits fatty acid amide hydrolase (FAAH ) in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

Subjects must:

* be healthy male subjects aged 18 to 45 years inclusive
* Have a body mass index (BMI) between 19 and 30 kg/m2 inclusive
* be able to provide a semen sample
* be willing to use an effective method of contraception (see Section 6.1) for the duration of the study and for 4 months after the last dose of study medication
* be able to comply with the requirements of the entire study
* give written informed consent

Exclusion Criteria:

Subjects must not:

* intend to father a child with their female partner or through sperm donation within 4 months after the last dose of study medication
* have had a vasectomy
* have a significant medical condition or a history of such a condition that the Investigator considers should exclude the subject from the study
* have multiple drug allergies or be allergic to any of the components of V158866 study medication or its matching placebo (see Section 7)
* have smoked more than 5 cigarettes per day in the 6 calendar months before study drug administration
* consume more than 28 units of alcohol per week, or have a significant history of alcohol abuse
* have a positive test for alcohol or drugs of abuse at screening or admission to any of the dosing sessions
* have donated blood or plasma in excess of 500 mL within 4 months before study drug administration
* have been exposed to any new investigational agent within 3 months before study drug administration
* have clinically relevant abnormal findings on vital signs
* have clinically significant abnormalities on laboratory screening tests
* have clinically relevant abnormal physical findings on examination
* have clinically relevant abnormal findings on 12-lead ECG
* have a mean QTc corrected using Bazett's correction (QTcB) at screening >430 msec (from 3 supine ECGs, performed at least 5 minutes apart)
* be seropositive for hepatitis B, hepatitis C or HIV viruses at screening
* have any medical or social reasons for not participating in the study raised by their General Practitioner/primary care physician
* have any other condition that might increase the risk to the individual or decrease the chance of obtaining satisfactory data, as assessed by the Investigator
* have had treatment with any prescription medicine within one month or any over-the-counter medicines, except for paracetamol, within one week before study drug administration

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of V158866 by assessing adverse events | Throughout the dosing phase with specific enquiries pre-dose and at 1, 2, 8, 24, 48 and 72 hours post-dose and at the post-study visit.
Evaluate the safety of V158866 by assessing vital signs | screen, Day -1, before and after each dose of V158866 or placebo (within 1 hour pre-dose and at 30 minutes (supine/semi-recumbent only), 1, 2, 3, 4, 8, 12, 24, 36, 48, 72 hours post-dose), post-study visit.
Evaluate the safety of V158866 by assessing ECGs | At screen, before and after each dose of V158866 or placebo (within 1 hour pre-dose and at 1, 2, 4, 8, 12, 24 and 72 hours post-dose), post-study visit.
Evaluate the safety of V158866 by assessing safety labs | At screen, Day 1, 24 hours and 72 hours after each dose of V158866 or placebo, and at the post-study visit.

SECONDARY OUTCOMES:
Blood concentration profile of V158866 | Samples will be collected within 15 minutes pre-dose and at 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48 and 72 hours after each dose
Measurement of FAAH activity and endocannabinoids | Up to 7 days post dosing

CONTACTS AND LOCATIONS:
Overall Officials: Steve Warrington, MD, Principal Investigator — Hammersmith Medicines Research Limited
Locations (1):
- Hammersmith Medicines Research Limited, London, United Kingdom